CLINICAL TRIAL: NCT05953753
Title: Impact and Process Evaluation of the Global Alliance for Improved Nutrition (GAIN) Enhancing Access to Safe and Nutritious Diets (ENSAND) Program in Nigeria
Brief Title: Enhancing Access to Safe and Nutritious Diets (ENSAND) Evaluation Nigeria
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The ENSAND project has been modified to focus on vegetable consumption in smallholder farmer households rather than egg consumption among children. The revisions are substantial enough to warrant closing this record and creating a new record.
Sponsor: RTI International (Other)
Collaborators: Datametrics Associates Ltd (Unknown); University of Nigeria Nsukka (Other); University of Abuja (Other)
Responsible Party: Principal Investigator, Valerie Flax, Senior Research Public Health Analyst, RTI International
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 424602
Record Dates: First submitted 2023-06-14; First posted 2023-07-20 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-02

CONDITIONS: Egg Consumption
Keywords: diet; eggs; market intervention; social and behavior change communication intervention; infants; children; Nigeria

STUDY DESIGN:
Intervention Model Description: Data will be collected through household surveys, value chain actor semi-structured interviews, KIIs, and FGDs. The protocol team has selected a subset of the intervention local government areas for the evaluation and identified an equal number of local government areas outside the program coverage area with similar characteristics to serve as the control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator)
  Interventions: Behavioral: Food system and demand generation
- Control/No intervention (No Intervention)

INTERVENTIONS:
Behavioral: Food system and demand generation — The project is focused on improving egg consumption through enhanced availability, accessibility, and improved demand. To achieve this goal, the project intervention mix will work through three pathways: access, enabling environment, and demand. The access pathway aims to sustain availability and consumption of eggs by school children (age 6-9 years) from BoP households through interventions targeted at the Poultry Association of Nigeria (PAN) and state lead egg aggregators for the HGSFP. The enabling environment pathway focuses on the broader institutional, governance, and political factors to support accessibility, availability, improved consumption, and increased consumer demand for eggs. The demand pathway will be addressed by mass media and interpersonal communication to increase the willingness and motivation of parents/caregivers in BoP households to support and sustain egg consumption by pre-school children in Kaduna State.
  Arms: Intervention

SUMMARY:
The Global Alliance for Improved Nutrition (GAIN) is implementing a program in 4 countries to increase consumption of healthy foods by improving supply, increasing demand, and improving the enabling environment for different targeted foods by operating at multiple levels - individuals, households, markets, producers, and policies. In Nigeria, the program is called Enhancing Access to Safe and Nutritious Diets (ENSAND). RTI and local partners propose to conduct impact and process evaluations of GAIN's program tailored to the theory of change and the target food for Nigeria. The evaluation in Nigeria will include a mix of quantitative and qualitative methods and will be guided by the RE-AIM (reach, effectiveness, adoption, implementation, and maintenance) evaluation framework.

DETAILED DESCRIPTION:
ENSAND seeks to increase the frequency of egg consumption among students in classes 1-3 in public primary schools and their younger siblings aged 6-59 months in local government areas (LGAs) with a high proportion of bottom of the pyramid (BoP) households. GAIN's intervention is two-pronged in Kaduna State. One component will involve improving the egg value chain supplying the Home-Grown School Feeding Program (HGSFP) for primary school children and the other will involve using a social marketing approach to increase parents' willingness to purchase and feed eggs to their young children aged 6-59 months. In Federal Capital Territory (FCT) and Kebbi States, GAIN's intervention will focus only on supplying eggs to primary school children.

This evaluation of the ENSAND program will use a parallel group mixed-methods quasi-experimental before-after design to assess the effectiveness of the intervention on children's frequency of egg consumption in Kaduna (intervention) and Kano (control) States. The evaluation will be carried out in 3 intervention and 3 control LGAs, with clustering at the level of the school. Data will be collected through household surveys with caregivers and school-aged children (N=1,332 at baseline and endline), egg value chain actor key informant interviews (KIIs, N=3) and semi-structured interviews (N=191) at baseline, midline, and endline, and focus group discussions (FGDs, N=9 FGDs at midline and endline) with caregivers of young children. Households with school- and pre-school aged children will be identified through the sampled public primary schools, and caregivers and school-aged children will be interviewed at baseline and endline in intervention and control LGAs. The same schools will be used at both times points but cross-sectional samples will be drawn at baseline and endline. Egg value chain actors will be identified in the intervention LGAs in Kaduna to participate in KIIs and semi-structured interviews at baseline, midline, and endline to assess changes in the functioning of the value chain over time. FGDs with caregivers of young children will be conducted at midline and endline. The qualitative findings will be used to understand experiences with the interventions and findings will be triangulated with results from the household and egg value chain interviews.

In FCT and Kebbi, the evaluation will be limited to KIIs (N=4) and semi-structured interviews (N=102) with egg value chain actors at baseline, midline, and endline. The findings will be used to validate and triangulate with the monitoring data GAIN will be collecting from value chain actors.

ELIGIBILITY:
Different populations will be targeted for different data collection methods. Eligibility criteria are detailed below for each data collection method.

Household Surveys

Inclusion Criteria:

* Adult caregiver who will be interviewed is 18 years or older;
* The household has a child in public primary school class 1-3 aged 6 - 9 years AND has a child 6-59 months
* The household earns <$3.20 per person per day;
* Able to speak English or Hausa;
* Provide informed consent to participate in the study.

Egg Value Chain Interviews

Inclusion Criteria:

* Be a PAN state manager, national or state HGSFP manager, poultry farmer, school-level HGSFP manager, health teacher, or egg retailer or wholesaler in the local government areas selected for the evaluation;
* Be 18 years or older;
* Able to speak English or Hausa;
* Provide informed consent to participate in the study.

Focus Group Discussions with Caregivers

Inclusion criteria:

* Caregivers with a child in class 1-3 and a child 6-59 months;
* Be 18 years or older;
* Able to speak English or Hausa;
* Provide informed consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1625 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Frequency of egg consumption by primary school children | Baseline (August 2023), Endline (August 2026) (3 years)
  Change in the mean frequency of egg consumption during the last 7 days by children in primary school classes 1-3 in BoP households
Frequency of egg consumption by pre-school children | Baseline (August 2023), Endline (August 2026) (3 years)
  Change in the mean frequency of egg consumption during the last 7 days by children 6-59 months in BoP households

SECONDARY OUTCOMES:
Frequency of egg purchase | Baseline (August 2023), Endline (August 2026) (3 years)
  Change in frequency of eggs purchased for children
Number of eggs purchased | Baseline (August 2023), Endline (August 2026) (3 years)
  Change in number of eggs purchased for children

CONTACTS AND LOCATIONS:
Overall Officials: Abiodun F Ipadeola, Principal Investigator — Datametrics Associates Ltd
Locations (1):
- Datametrics Associates Ltd., Abuja, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Dataset will be shared through Nesstar.